CLINICAL TRIAL: NCT04505462
Title: Short-Term Effects of Therapeutic Diet in Dialysis Patients
Brief Title: Dietary Therapy in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wan-Chuan Tsai, Principal Investigator, Assistant Professor, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FEMH-IRB-109112-F
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Therapeutic diet; Mineral metabolism; Uremic toxins; Inflammation; Immune; End-stage kidney disease
MeSH Terms: conditions — Inflammation; Kidney Failure, Chronic | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: A randomized, active-controlled trial with cross-over design
Who Masked: Outcomes Assessor
Masking Description: Laboratory technicians who assess the study outcomes will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study diet (Experimental): 7-day therapeutic diet intervention as experimental group
  Interventions: Other: Therapeutic diet
- Usual diet (No Intervention): 7-day usual diet as control group, no dietary intervention in this group, participants consumed their habitual diet

INTERVENTIONS:
Other: Therapeutic diet — A special healthy diet for dialysis patients
  Other Names: Dietary therapy
  Arms: Study diet

SUMMARY:
Patients with end-stage kidney disease have hyperphosphatemia and accumulated uremic toxin level due to decreased urine excretion ability. Unhealthy diet causes altered mineral metabolism, elevated uremic toxin level, immune dysregulation, and inflammation. The investigators hypothesize that therapeutic diet intervention reverses altered mineral metabolism, elevated uremic toxin level, immune dysregulation, and inflammation. In this study, the investigators crafted 7-day special healthy diet to illustrate the clinical implications of therapeutic diet for dialysis patients.

DETAILED DESCRIPTION:
The risk of cardiovascular disease (CVD) and mortality in patients with end-stage kidney disease (ESKD) is far greater than those in the general population. Emerging evidence suggests that unhealthy diet causes altered mineral metabolism, disturbance of gut microbiota (dysbiosis) with elevated uremic toxin level, immune dysregulation, and inflammation; these abnormalities are strongly related to development of CVD. Little is known about the relationship between therapeutic diet intervention and cardiovascular risk in patients with ESKD. Recently, the study of the investigators showed that ESKD patients undergoing hemodialysis who consumed very low-phosphate diet, phosphate-to-protein ratio (PPR) value of 8 mg/g, experienced an extra reduction of serum phosphorus level by 0.61 mg/dL compared with that of low-phosphate diet, PPR value of 10 mg/g.

The aim of the study is to explore the effect of 7-day therapeutic diet intervention on changes of altered mineral metabolism, uremic toxin production, immune dysregulation and inflammation, highlighting the important role of dietary modification in dialysis population.

It is to conduct a randomized controlled trial with cross-over design at a hemodialysis unit of tertiary teaching hospital in Northern Taiwan. Subjects with aged older than 20 years, ESKD undergoing maintenance dialysis for more than three months, having adequate dialysis and serum intact parathyroid hormone less than 800 pg/mL will be included. Participants will be randomly assigned into two groups: those in group A will receive study diet for 7 days, followed by 4-week washout period and then receive 7-day usual diet. The opposite order of diets will be prescribed in group B. The study meals are prepared in the hospital cafeteria. Dietary compositions of the study diets were analyzed before the start of the study. The study outcome measures are difference in change-from-baseline values of altered mineral metabolism, uremic toxin production, immune dysregulation and inflammation between the therapeutic diet and the usual diet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with aged older than 20 years, ESKD undergoing maintenance dialysis for more than three months, having adequate dialysis, serum intact parathyroid hormone less than 800 pg/mL and good dietary compliance

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from the study:

  1. Serum albumin level less than 2.5 g/dL
  2. Hospitalization within the past 4 weeks
  3. Prebiotics, probiotics, symbiotics or antibiotics use within the past 4 weeks
  4. History of psychiatric disorders
  5. Having mental retardation
  6. Those who dislike of the study meals
  7. Soft diet requirement
  8. Vegetarian

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Concentrations of intact fibroblast growth factor 23 (pg/mL) | 7 days
  Difference in change-from-baseline intact fibroblast growth factor 23 (pg/mL) between therapeutic diet and usual diet

SECONDARY OUTCOMES:
Concentrations of C-terminal fibroblast growth factor 23 (RU/mL) | 7 days
  Difference in change-from-baseline C-terminal fibroblast growth factor 23 (RU/mL) between therapeutic diet and usual diet
Concentrations of phosphate (mg/dL) | 7 days
  Difference in change-from-baseline phosphate (mg/dL) between therapeutic diet and usual diet
Concentrations of calcium (mg/dL) | 7 days
  Difference in change-from-baseline calcium (mg/dL) between therapeutic diet and usual diet
Concentrations of intact parathyroid hormone (pg/mL) | 7 days
  Difference in change-from-baseline intact parathyroid hormone (pg/mL) between therapeutic diet and usual diet
Concentrations of free indoxyl sulfate (mg/L) | 7 days
  Difference in change-from-baseline free indoxyl sulfate (mg/L) between therapeutic diet and usual diet
Concentrations of free p-cresol sulfate (mg/L) | 7 days
  Difference in change-from-baseline free p-cresol sulfate (mg/L) between therapeutic diet and usual diet
Concentrations of pre-albumin (g/dL) | 7 days
  Difference in change-from-baseline pre-albumin (g/dL) between therapeutic diet and usual diet
Concentrations of albumin (g/dL) | 7 days
  Difference in change-from-baseline albumin (g/dL) between therapeutic diet and usual diet
Concentrations of C-reactive protein (mg/dL) | 7 days
  Difference in change-from-baseline C-reactive protein (mg/dL) between therapeutic diet and usual diet
Absolute number (per μl blood) of CD4+ (cluster of differentiation 4) T cells | 7 days
  Difference in change-from-baseline absolute number (per μl blood) of CD4+ T cells between therapeutic diet and usual diet
Absolute number (per μl blood) of CD8+ (cluster of differentiation 8) T cells | 7 days
  Difference in change-from-baseline absolute number (per μl blood) of CD8+ T cells between therapeutic diet and usual diet
Absolute number (per μl blood) of monocytes | 7 days
  Difference in change-from-baseline absolute number (per μl blood) of monocytes between therapeutic diet and usual diet
Percentage (%) of CD4+ (cluster of differentiation 4) T cells | 7 days
  Difference in change-from-baseline percentage (%) of CD4+ (cluster of differentiation 4) T cells between therapeutic diet and usual diet
Percentage (%) of CD8+ (cluster of differentiation 8) T cells | 7 days
  Difference in change-from-baseline percentage (%) of CD8+ (cluster of differentiation 8) T cells between therapeutic diet and usual diet
Percentage (%) of monocytes | 7 days
  Difference in change-from-baseline percentage (%) of monocytes between therapeutic diet and usual diet

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Chuan Tsai, M.D., Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual-level deidentified participant data will be made available by the corresponding author of the paper upon request by email. The data will be available for 3 years after formal publication.
Supporting Information: Study Protocol
Time Frame: The data will become available after completing the study for 1 year and for 3 years after formal publication.
Access Criteria: Data will be made available by the corresponding author of the paper upon request by email.

REFERENCES:
- [Background] Tsai WC, Wu HY, Peng YS, Hsu SP, Chiu YL, Yang JY, Chen HY, Pai MF, Lin WY, Hung KY, Chu FY, Tsai SM, Chien KL. Short-Term Effects of Very-Low-Phosphate and Low-Phosphate Diets on Fibroblast Growth Factor 23 in Hemodialysis Patients: A Randomized Crossover Trial. Clin J Am Soc Nephrol. 2019 Oct 7;14(10):1475-1483. doi: 10.2215/CJN.04250419. Epub 2019 Sep 13. PMID 31519550
- [Background] Tsai WC, Wu HY, Peng YS, Hsu SP, Chiu YL, Chen HY, Yang JY, Ko MJ, Pai MF, Tu YK, Hung KY, Chien KL. Effects of lower versus higher phosphate diets on fibroblast growth factor-23 levels in patients with chronic kidney disease: a systematic review and meta-analysis. Nephrol Dial Transplant. 2018 Nov 1;33(11):1977-1983. doi: 10.1093/ndt/gfy005. PMID 29420827
- [Derived] Tsai WC, Hsu SP, Chiu YL, Wu HY, Luan CC, Yang JY, Pai MF, Lin CJ, Lin WY, Sun WH, Peng YS. Short-Term Effects of a Therapeutic Diet on Biochemical Parameters in Hemodialysis Patients: A Randomized Crossover Trial. J Ren Nutr. 2023 Nov;33(6):731-739. doi: 10.1053/j.jrn.2023.04.003. Epub 2023 Apr 27. PMID 37120127